CLINICAL TRIAL: NCT07192185
Title: Systemic Chemotherapy With FOLFOX Plus Atezolizumab & Bevacizumab for Patients With Advanced HCC Who Previously Received Atezolizumab & Bevacizumab: a Single Arm Trial.
Brief Title: Systemic Chemotherapy With FOLFOX Plus Atezolizumab & Bevacizumab for Patients With Advanced HCC Who Previously Received Atezolizumab & Bevacizumab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOLFOX+TA as 2nd treatment
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: FOLFOX; Atezolizumab plus bevacizumab; Systemic chemotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Folfox protocol; atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOLFOX+TA (Experimental): Systemic chemotherapy with FOLFOX plus Atezolizumab & bevacizumab
  Interventions: Drug: FOLFOX; Drug: Atezolizumab & Bevacizumab

INTERVENTIONS:
Drug: FOLFOX — oxaliplatin 85mg/m2 + leucovorin 400mg/m2 + 5-fu 400mg/m2 + 5-fu 2400mg/m2 46h iv.drip Q3W
Drug: Atezolizumab & Bevacizumab — Atezolizumab 1200mg iv.drip + Bevacizumab 15mg/kg iv.drip Q3w

SUMMARY:
Atezolizumab plus bevacizumab is the first-line treatment for advanced hepatocellular carcinoma (HCC). However, the effect of the second-line treatment after the progress of Atezolizumab plus bevacizumab therapy remains unsatisfactory. This is a prospective trial to investigate the efficacy and safety of systemic chemotherapy with FOLFOX plus Atezolizumab & bevacizumab as second-line treatment for patients with advanced HCC who previously received atezolizumab plus bevacizumab

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* Barcelona clinic liver cancer-stage C
* Patients who have previously received first-line treatment with atezolizumab plus bevacizumab and who have shown tumor progression as confirmed by imaging studies. No other systemic treatments have been administered.
* Eastern Cooperative Oncology Group performance status of 0 to 2
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* The following laboratory parameters:

Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 30 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3

• Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
ORR via mRECIST | 12 months
  CR+PR via mRECIST

SECONDARY OUTCOMES:
OS | 12 months
  overall survival was defined as the duration from the date of randomization until the date of death from any cause. Participants who were lost to follow-up were censored at the last date the participant was known to be alive, and participants who remained alive were censored at the time of data cutoff.
Progression Free Survival (PFS) | 12 months
  PFS was defined as the time from the date of randomization to the date of first documentation of disease progression based on modified Response Evaluation Criteria in Solid Tumors (mRECIST), or date of death, whichever occurred first.
Adverse Events | 12 months
  Number of adverse events. Postoperative adverse events were graded based on CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China